

# **Clinical Trial Protocol**

| | Document Number: | c24401085-02 |
|---|---|---|
| EudraCT No. | 2018-002792-18 | |
| BI Trial No. | 1405-0007 | |
| BI Investigational<br>Medicinal Product | BI 1323495 | |
| Title | Relative bioavailability of BI 1323495 following oral administration under fed and fasted conditions in healthy male subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study) | |
| Lay Title | A study to test how food influences the amount of BI 1323495 in the blood of healthy men | |
| Clinical Phase | I | |
| Trial Clinical<br>Monitor | Phone: | |
| Principal Investigator | Fax: | |
| | Phone:<br>Fax: | |
| Status | Final Protocol (Revised Protocol (based on global amendment 1)) | |
| Version and Date | Version: 2.0 | Date: 22 November 2018 |

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

**Trial Protocol** 

**** 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Company name | Boehringer Ingelheim |
|---|---|
| Protocol date | 1 August 2018 |
| Revision date | 22 November 2018 |
| BI trial number | 1405-0007 |
| Title of trial | Relative bioavailability of BI 1323495 following oral administration under fed and fasted conditions in healthy male subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study) |
| Principal Investigator | |
| Trial site | |
| Clinical phase | I |
| Trial rationale | This food interaction study will generate pharmacokinetic information under fed conditions versus the fasted state to support the future development in patients. |
| Trial objective | To investigate the relative bioavailability of a single oral dose of BI 1323495 under fed and fasted conditions |
| Trial design | Randomised, open-label, two-way crossover design |
| Trial endpoints | Primary endpoints: AUC $_{0-tz}$ and C $_{max}$ of BI 1323495<br>Secondary endpoints: AUC $_{0-\infty}$ of BI 1323495 |
| Number of subjects | |
| total entered | 12 |
| each treatment | 12 |
| Diagnosis | Not applicable |
| Main criteria<br>for inclusion | Healthy male subjects, age of 18 to 45 years (inclusive), body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive) |
| Test product | BI 1323495 tablet formulation |
| dose<br>mode of admin. | Oral with 240 mL of water following a high fat, high calorie meal (treatment test (T)) and after an overnight fast of at least 10 h (treatment reference (R)) |

**22 November 2018** 

c24401085-02 Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Duration of treatment | One day (single dose) for each treatment |
|---|---|
| Statistical methods | Relative bioavailability will be estimated by the ratios of the geometric means (test/reference) for the primary and secondary endpoints. Additionally, their two-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at a 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified. The statistical model will be an analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period and treatment. CIs will be calculated based on the residual error from the ANOVA. Descriptive statistics will be calculated for all endpoints. |

**22 November 2018** 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

**FLOW CHART** 

c24401085-02


c24401085-02 Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **TABLE OF CONTENTS**

| TI | LLE I | PAGE | 1 |
|---|---|---|---|
| CL | INIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| FL | ow ( | CHART | 4 |
| | | OF CONTENTS | |
| | | VIATIONS | |
| 1. | | RODUCTION | |
| | 1.1 | MEDICAL BACKGROUND | |
| | 1.2 | DRUG PROFILE | 12 |
| | | 1.2.4 Clinical experience in humans | |
| | | 1.2.4.1 Clinical experience with BI 1323495 | 14 |
| | | 1.2.5 Residual Effect Period | 19 |
| | 1.3 | RATIONALE FOR PERFORMING THE TRIAL | |
| | 1.4 | BENEFIT - RISK ASSESSMENT | |
| 2. | | AL OBJECTIVES AND ENDPOINTS | |
| | 2.1 | MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS | |
| | 2.1 | 2.1.1 Main objectives | |
| | | 2.1.2 Primary endpoints | |
| | | 2.1.3 Secondary endpoint | |
| 3. | DES | SCRIPTION OF DESIGN AND TRIAL POPULATION | . 24 |
| | 3.1 | OVERALL TRIAL DESIGN AND PLAN | 24 |
| | 3.2 | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUPS | 24 |
| | 3.3 | SELECTION OF TRIAL POPULATION | 24 |
| | | 3.3.1 Main diagnosis for trial entry | |
| | | 3.3.2 Inclusion criteria | |
| | | 3.3.3 Exclusion criteria | |
| | | 3.3.4 Withdrawal of subjects from treatment or assessments | <b>26</b> |
| | | 3 3 4 1 Discontinuation of trial freatment | ブル |

5.2

5.2.1

5.2.2

#### c24401085-02 Trial Protocol

**** 

| Pı | oprietary | confidential i | information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated con | mpanies |
|---|---|---|---|---|
| | | | 3.3.4.2 Withdrawal of consent to trial participation | 27 |
| | | | 3.3.4.3 Discontinuation of the trial by the sponsor | |
| | | 3.3.5 | Replacement of subjects | |
| 4. | TRI | EATMI | ENTS | |
| | 4.1 | | STIGATIONAL TREATMENTS | |
| | | 4.1.1 | Identity of the Investigational Medicinal Products | |
| | | 4.1.2 | Selection of doses in the trial and dose modifications | |
| | | 4.1.3 | Method of assigning subjects to treatment groups | 30 |
| | | 4.1.4 | Drug assignment and administration of doses for each subje | |
| | | 4.1.5 | Blinding and procedures for unblinding | 31 |
| | | 4.1.6 | Packaging, labelling, and re-supply | 31 |
| | | 4.1.7 | Storage conditions | 32 |
| | | 4.1.8 | Drug accountability | 32 |
| | 4.2 | | ER TREATMENTS, EMERGENCY PROCEDURES, | |
| | | REST | RICTIONS | |
| | | 4.2.1 | Other treatments and emergency procedures | 32 |
| | | 4.2.2 | Restrictions | |
| | | | 4.2.2.1 Restrictions regarding concomitant treatment | |
| | | | 4.2.2.2 Restrictions on diet and life style | |
| | 4.3 | TREA | TMENT COMPLIANCE | 33 |
| <b>5.</b> | ASS | ESSM | ENTS | 34 |
| | 5.1 | ASSES | SSMENT OF SAFETY | 34 |
| | | 5.1.1 | Physical examination | 34 |
| | | 5.1.2 | Vital signs | |
| | | 5.1.3 | Safety laboratory parameters | 34 |
| | | 5.1.4 | Electrocardiogram | 37 |
| | | 5.1.5 | Assessment of adverse events | 37 |
| | | | 5.1.5.1 Definitions of adverse events | 37 |

 5.1.5.1.1 Adverse event
 37

 5.1.5.1.2 Serious adverse event
 38

 5.1.5.1.3 AEs considered 'Always Serious'
 38

 5.1.5.1.4 Adverse events of special interest
 39

 5.1.5.1.5 Intensity (severity) of AEs
 39

 5.1.5.1.6 Causal relationship of AEs
 39

 5.1.5.2.1 AE collection
 40

 5.1.5.2.2 AE reporting to the sponsor and timelines
 41

 5.1.5.2.3 Information required
 41

 5.1.5.2.4 Pregnancy
 41

5.1.5.2 Adverse event collection and reporting .......40

Assessment of pharmacokinetics ......42

Methods of sample collection ......42

PHARMACOKINETICS.......42

DRUG CONCENTRATION MEASUREMENTS AND

c24401085-02 Trial Protocol 

| _ | - | | | | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dec | amatam | , aantidantia | linformatio | $\sim$ $\sim$ $\sim$ $\sim$ $\sim$ $\sim$ | oohringer I | naalhaim | Intornational | Combu or | one or more of it | a affiliated as | manning |
| FIO | пістагу | COHITAGILIA | і шпоппацо | $\mathbf{n} \otimes \mathbf{z} \mathbf{o} \mathbf{n}$ | ochinisci n | usemenn | пистнанопат | CHIRDLE OF C | one or more or it | s arrinateu cu | minames |

| | | 5.2.2.1 Blood sampling for pharmacokinetic analysis | 42 |
|---|---|---|---|
| | | 5.2.3 Analytical determinations | |
| | | 5.2.4 Pharmacokinetic - pharmacodynamic relationship | |
| | 5.3 | BIOBANKING | |
| | 5.4 | OTHER ASSESSMENTS | |
| | 5.5 | APPROPRIATENESS OF MEASUREMENTS | 43 |
| 6. | INV | ESTIGATIONAL PLAN | 44 |
| | 6.1 | VISIT SCHEDULE | |
| | 6.2 | DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS | |
| | | 6.2.1 Screening | 44 |
| | | 6.2.2 Treatment periods | |
| | | 6.2.3 Follow-up period and trial completion | 45 |
| 7. | STA | ATISTICAL METHODS AND DETERMINATION OF | |
| | SAN | MPLE SIZE | 46 |
| | 7.1 | STATISTICAL DESIGN – MODEL | 4 <mark>6</mark> |
| | 7.2 | NULL AND ALTERNATIVE HYPOTHESES | 46 |
| | 7.3 | PLANNED ANALYSES | 46 |
| | | 7.3.1 Primary endpoint analyses | 47 |
| | | 7.3.2 Secondary endnoint analyses | 48 |
| | | 7.3.4 Safety analyses | 49 |
| | 7.4 | INTERIM ANALYSES | |
| | 7.5 | HANDLING OF MISSING DATA | |
| | | 7.5.1 Safety | 50 |
| | | 7.5.2 Pharmacokinetics | 50 |
| | 7.6 | RANDOMISATION | |
| | 7.7 | DETERMINATION OF SAMPLE SIZE | 50 |
| 8. | INF | ORMED CONSENT, TRIAL RECORDS, DATA | |
| | PRO | OTECTION, PUBLICATION POLICY, AND | |
| | AD | MINISTRATIVE STRUCTURE | <u>51</u> |
| | 8.1 | TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED | |
| | | CONSENT | 51 |
| | 8.2 | DATA QUALITY ASSURANCE | 52 |
| | 8.3 | RECORDS | 52 |
| | | 8.3.1 Source documents | |
| | | 8.3.2 Direct access to source data and documents | |
| | | 8.3.3 Storage period of records | |
| | 8.4 | EXPEDITED REPORTING OF ADVERSE EVENTS | |
| | 8.5 | STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY | Y54 |

**22 November 2018** 

| 24401085-02 | Trial Protocol | Page 8 of 6 |
|---|---|---|
| Proprietary confidential inform | nation © 2018 Boehringer Ingelheim Internationa | l GmbH or one or more of its affiliated companies |

| | | 8.5.1 Collection, storage and future use of biological samples a | ınd |
|---|---|---|---|
| | | corresponding data | 54 |
| | 8.6 | TRIAL MILESTONES | 54 |
| | <b>8.7</b> | ADMINISTRATIVE STRUCTURE OF THE TRIAL | 55 |
| 9. | REF | ERENCES | 56 |
| | 9.1 | PUBLISHED REFERENCES | 56 |
| | 9.2 | UNPUBLISHED REFERENCES | 58 |
| 10. | APP | ENDICES | 59 |
| 11. | DES | CRIPTION OF GLOBAL AMENDMENT(S) | 60 |
| | | GLOBAL AMENDMENT 1 | |

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ABBREVIATIONS**

ADME Absorption, distribution, metabolism, and excretion

AE Adverse event

AESI Adverse events of special interest

ANOVA Analysis of variance

AUC $_{0-\infty}$  Area under the concentration-time curve of the analyte in plasma over the

time interval from 0 extrapolated to infinity

 $AUC_{0-tz}$  Area under the concentration-time curve of the analyte in plasma over the

time interval from 0 to the last quantifiable data point

BI Boehringer Ingelheim

BMI Body mass index (weight divided by height squared)

BP Blood pressure

CA Competent authority

CI Confidence interval

C<sub>max</sub> Maximum measured concentration of the analyte in plasma

CML Clinical Monitor Local

CRF Case Report Form, paper or electronic (sometimes referred to as 'eCRF')

CTP Clinical trial protocol
CTR Clinical trial report

DILI Drug induced liver injury

ECG Electrocardiogram

eCRF Electronic case report form eDC Electronic data capture

EDTA Ethylenediaminetetraacetic acid

EoTrial End of trial

EudraCT European Clinical Trials Database

FU Follow-up

GCP Good Clinical Practice

**22 November 2018** 

Boehringer Ingelheim BI Trial No.: 1405-0007

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

HR Heart rate

IB Investigator's brochure

IC<sub>50</sub> Half-maximal inhibitory concentration

IEC Independent Ethics CommitteeIPV Important protocol violationIRB Institutional Review Board

ISF Investigator site file

LC-MS/MS Liquid chromatography with tandem mass spectrometry

MDA Methylenedioxyamphetamine
MDMA Methylenedioxymethamphetamine

MedDRA Medical Dictionary for Regulatory Activities

NOAEL No observed adverse effect level

PKS Pharmacokinetic(s)
PKS Pharmacokinetic set

PR Pulse rate

QT Time between start of the Q-wave and the end of the T-wave in an

electrocardiogram

QT or QT interval corrected for heart rate using the method of Fridericia (QTcF)

or Bazett (QTcB)

R Reference treatment
REP Residual effect period
SAE Serious adverse event

SCR Screening

SOP Standard operating procedure T Test product or treatment

TS Treated set

TSAP Trial statistical analysis plan

ULN Upper limit of normal

XTC Ecstasy

**22 November 2018** 

c24401085-02 Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. INTRODUCTION

This trial will investigate the effect of food on pharmacokinetics of BI 1323495.

# 1.1 MEDICAL BACKGROUND

c24401085-02

**22 November 2018** 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

#### 1.2 **DRUG PROFILE**


c24401085-02

**22 November 2018** 

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Boehringer Ingelheim BI Trial No.: 1405-0007 c24401085-02

**22 November 2018** 

Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For a more detailed description of the BI 1323495 profile, please refer to the current Investigator's Brochure (IB) (c21238478-01).

# 1.2.4 Clinical experience in humans

#### 1.2.4.1 Clinical experience with BI 1323495

At the time of CTA submission of this trial, the first in man study 1405-0001 had been initiated. This partially randomized within dose groups, placebo-controlled trial investigates the safety, tolerability, pharmacokinetics and pharmacodynamics of single rising oral doses of BI 1323495 as tablet formulation. As of 14 November 2018, the clinical part has been completed as planned. A total of 63 subjects were randomized to treatment with either

c24401085-02 Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

placebo (N=15) or single ascending doses of

BI 1323495 (N=6 per dose). An overview on preliminary results of this trial is given in the following.

Treatments with BI 1323495 tablets or placebo were safe and well tolerated at all doses investigated. Overall, 16 out of 48 subjects treated with BI 1323495 (33.3%) and 2 out of 15 subjects treated with placebo (13.3%) were reported with at least 1 AE following drug administration. No dose dependency was observed for the different BI 1323495 treatment groups. The most frequently reported AE was headache, observed in 6 subjects (12.5%) dosed with BI 1323495 and 2 subjects (13.3%) on placebo. The incidence of headache appeared similar between the different BI 1323495 dose groups and placebo.

AEs were generally of short duration and mild in intensity apart from 1 case of moderate headache moderate common cold reported by one subject , and 1 case of moderate rhinitis . Severe or serious AEs were not reported. All AEs were followed-up until resolved.

A summary of AEs reported following study drug treatment is shown in Table 1.2.4.1: 1.

Table 1.2.4.1: 1 Number (percentage) of subjects with AEs following administration of BI 1323495 or placebo in SRD trial 1405-0001

| AE reported | Placebo | | | | BI 1323495 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| term | | | | | | | | | | Total BI |
| | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| No. of subjects | 15<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 6<br>(100.0) | 48<br>(100.0) |
| Total with on treatment AEs | 2 (13.3) | 3 (50.0) | 2 (33.3) | 1 (16.7) | 2 (33.3) | 1 (16.7) | 2 (33.3) | 3 (50.0) | 2 (33.3) | 16<br>(33.3) |
| Headache | 2 (13.3) | 3 (50.0) | 1 (16.7) | - | - | - | - | 1 (16.7) | 1 (16.7) | 6 (12.5) |
| Tiredness | - | - | - | 1 (16.7) | 1 (16.7) | - | - | | - | 2 (4.2) |
| Diarrhoea | - | - | 1 (16.7) | - | - | - | - | 1 (16.7) | - | 2 (4.2) |
| Stiff neck | - | - | - | - | 1 (16.7) | - | - | | - | 1 (2.1) |
| Malaise | - | - | - | - | - | 1 (16.7) | - | | - | 1 (2.1) |
| Common cold | - | - | - | - | - | - | 1 (16.7) | - | - | 1 (2.1) |
| Improved breathing | _ | - | - | - | - | - | - | 1 (16.7) | - | 1 (2.1) |
| ALT increase | - | - | - | - | - | - | 1 (16.7) | - | - | 1 (2.1) |
| GLDH increase | - | - | - | - | - | - | 1 (16.7) | - | - | 1 (2.1) |
| Rhinitis | - | - | - | - | - | - | - | - | 1<br>(16.79 | 1 (2.1) |

Clinically relevant changes in ECGs, vital signs (BP, pulse) or safety laboratory parameters were to be reported as adverse events.

**22 November 2018** 

c24401085-02 Trial Protocol Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

No adverse events based on ECG or vital signs were reported. Also no trends of changes were observed.

Noteworthy: Subject (BI 1323495) presented with an increase in pulse rate compared to baseline from 5h to 12h postdose, i.e. after the end of bed rest period. Systolic blood pressure showed also a trend to higher values in the same period. This is explained by increased physical activity and not considered as clinically relevant. Furthermore, subject who was randomised to placebo, had single ECGs with absolute QT of 502 ms (2/3 ECGs at 2h p.a.) and 500 ms (1/3 ECGs at 3h p.a.). Change from baseline was below 60 ms and QTc below 430 ms.

The clinical laboratory evaluation included the analysis of haematology, coagulation, enzymes, substrates, electrolytes, urinalysis, and inflammatory parameters. In general, values of measured laboratory parameters were within or only slightly outside the respective reference ranges. There were no hints for relevant changes over time and no relevant differences between the treatment groups (including placebo) in any of the safety laboratory parameters measured.

Noteworthy: Subject (BI 1323495) presented with mild elevation of ALT and GLDH. Highest value for ALT was seen 4 days after drug administration (96 U/L, ULN=50 U/L); follow-up measurements were done until returned to almost normalized value of 51 U/L at 16 days postdose. Highest value for GLDH was already seen at 4h p.a. (11 U/L, ULN= 7.0 U/L). GLDH value returned to normal range 5 days after drug administration. Both laboratory findings are reported as adverse events of mild intensity and potentially related to the administration of BI 1323495.

#### Pharmacokinetic results:

Plasma samples were taken up to 96 h after drug administration. Preliminary PK data analysis for BI 1323495 used planned vs actual sampling times for all dose groups. Bioanalytical data of BI 1323495 and PK calculation is preliminary and subject to change.

c24401085-02

**22 November 2018** 

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c24401085-02

**22 November 2018** 

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c24401085-02


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1.2.5 Residual Effect Period

The Residual Effect Period (REP) of BI 1323495, i.e., the time interval when measurable drug levels or PD effects are still likely to be present after administration, is not yet known. Therefore, all AEs with an onset between start of treatment and the end of trial examination (last per protocol contact) will be considered on treatment.

#### 1.3 RATIONALE FOR PERFORMING THE TRIAL

In the ongoing single rising dose study, only pharmacokinetic data under fasted conditions are investigated for BI 1323495. The planned food interaction study will generate pharmacokinetic information under fed conditions to support the future development in patients.

#### 1.4 BENEFIT - RISK ASSESSMENT

Participation in this clinical trial is without any (therapeutic) benefit for healthy subjects. Their participation, however, is of major importance for the development of a new orally available drug, which might improve the therapy in patients with COPD and emphysema. The subjects are exposed to the risks of the study procedures and the risks related to the exposure to the trial medication.

#### Procedure-related risks

The use of an indwelling venous catheter or venepuncture for e.g. blood sampling may result in mild bruising, and in rare cases, in transient inflammation of the wall of the vein, or nerve injury, potentially resulting in paraesthesia, reduced sensibility, and/or pain for an indefinite period.

The total volume of blood withdrawn per subject during the entire study will not exceed the volume of a normal blood donation (500 mL). No health-related risk to healthy subjects is expected from withdrawal of this volume of blood.

Drug-related risks and safety measures

c24401085-02

**22 November 2018** 

Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**22 November 2018** 

C24401085-02 Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In this food effect trial, subjects will receive two single doses of once under fasted and once under fed conditions. Administration of BI 1323495 under fed conditions may cause an increase of plasma concentrations of BI 1323495. However, based on modelling data for the tablet formulation used in the SRD trial and this food effect trial only a minimal food effect is expected for a dose of resulting in plasma concentrations below those exposures seen in the SRD trial following doses of and above.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 2. TRIAL OBJECTIVES AND ENDPOINTS

#### 2.1 MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS

#### 2.1.1 Main objectives

The main objective of this trial is to assess the effect of food on the pharmacokinetics of an oral tablet formulation of BI 1323495 by investigating the relative bioavailability following single dose administration under fed and fasted conditions.

#### 2.1.2 Primary endpoints

The following pharmacokinetic parameters will be determined for BI 1323495:

- AUC<sub>0-tz</sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- C<sub>max</sub> (maximum measured concentration of the analyte in plasma)

# 2.1.3 Secondary endpoint

The following pharmacokinetic parameter will be determined for BI 1323495:

• AUC<sub>0- $\infty$ </sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)

c24401085-02

**22 November 2018** 

Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

# 3.1 OVERALL TRIAL DESIGN AND PLAN

The study will be performed as a randomised, open-label, two-way crossover trial in healthy male subjects in order to compare the test treatment (T) to the reference treatment (R). The treatments will be two single oral doses of BI 1323495 separated by a washout period between the treatments:

Treatment T: tablets of BI 1323495, <u>fed</u>
Treatment R: tablets of BI 1323495, fasted

The subjects will be randomly allocated to the 2 treatment sequences (T-R or R-T). For details, refer to Section 4.1.

An overview of all relevant trial activities is provided in the <u>Flow Chart</u>. For visit schedule and details of trial procedures at selected visits, refer to Sections <u>6.1</u> and <u>6.2</u>, respectively.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUPS

For relative bioavailability trials, the crossover design is preferred because of its efficiency: since each subject serves as his own control, the comparison between treatments is based on an intra-subject comparison, thus removing inter-subject variability from the comparison between treatments (R94-1529).

The open-label treatment is not expected to bias results, since the study endpoints are derived from measurement of plasma concentrations of the analyte, which are provided by a bioanalytical laboratory that is blinded to treatment allocation.

#### 3.3 SELECTION OF TRIAL POPULATION

It is planned that 12 healthy male subjects will enter the study. They will be recruited from the volunteers' pool of the trial site.

Only male subjects will be included in the study because no data on reproductive toxicology are available at this time.

A log of all subjects enrolled into the trial (i.e. who have signed informed consent) will be maintained in the ISF irrespective of whether they have been treated with investigational drug or not.

#### 3.3.1 Main diagnosis for trial entry

The study will be performed in healthy subjects.

## 3.3.2 Inclusion criteria

Subjects will only be included in the trial if they meet the following criteria:

**22 November 2018** 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
- 2. Age of 18 to 45 years (inclusive)
- 3. BMI of 18.5 to  $29.9 \text{ kg/m}^2$  (inclusive)
- 4. Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

#### 3.3.3 Exclusion criteria

Subjects will not be allowed to participate, if any of the following general criteria apply:

- 1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
- 2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
- 3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
- 4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
- 5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
- 6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
- 7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
- 8. History of relevant orthostatic hypotension, fainting spells, or blackouts
- 9. Chronic or relevant acute infections
- 10. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
- 11. Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
- 12. Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
- 13. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
- 14. Inability to refrain from smoking on specified trial days
- 15. Alcohol abuse (consumption of more than 30 g per day)
- 16. Drug abuse or positive drug screening
- 17. Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial

Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 18. Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
- 19. Inability to comply with the dietary regimen of the trial site
- 20. A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are greater than 450 ms, if confirmed by a 2nd ECG recording) or any other relevant ECG finding at screening
- 21. A history of additional risk factors for *Torsade de Pointes* (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
- 22. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
- 23. Subjects with female partner of childbearing potential who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial
- 24. Current or history of relevant kidney, urinary tract diseases or abnormalities (e.g. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure)
- 25. Estimated glomerular filtration rate according to CKD-EPI formula < 90 mL/min at screening
- 26. Within 10 days prior to administration of trial medication, use of any drug that could reasonably inhibit platelet aggregation or coagulation (e.g., acetylsalicylic acid)
- 27. Liver enzyme (ALT, AST, GGT) values above upper limit of normal at the screening examination

For study restrictions, refer to Section <u>4.2.2</u>.

# 3.3.4 Withdrawal of subjects from treatment or assessments

Subjects may discontinue trial treatment or withdraw consent to trial participation as a whole ('withdrawal of consent') with very different implications; please see Sections 3.3.4.1 and 3.3.4.2 below.

If a subject is removed from or withdraws from the trial prior to the first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after the first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF; in addition, the data will be included in the CRF and will be reported in the CTR. At the time of discontinuation, a complete end of trial examination will be performed, if possible, and the information will be recorded in the CRF. If the discontinuation occurs before the end of the REP (see Section 1.2.5), the discontinued subject should if possible be questioned for AEs and concomitant therapies at or after the end of the REP in order to ensure collection of AEs and concomitant therapies throughout the REP, if not contrary to any consent withdrawal of the subject.

c24401085-02

Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.4.1 Discontinuation of trial treatment

An individual subject will discontinue trial treatment if:

- 1. The subject wants to discontinue trial treatment, without the need to justify the decision
- 2. The subject has repeatedly shown to be non-compliant with important trial procedures and, in the opinion of both, the investigator and sponsor representative, is not willing or able to adhere to the trial requirements in the future.
- 3. The subject needs to take concomitant medication that interferes with the investigational medicinal product or other trial treatment
- 4. The subject can no longer receive trial treatment for medical reasons (such as surgery, adverse events [AEs], or diseases)
- 5. The subject has an elevation of AST and/or ALT ≥3-fold upper limit of normal (ULN) and an elevation of total bilirubin ≥2-fold ULN (measured in the same blood sample) and/or needs to be followed up according to the DILI checklist provided in the ISF.
- 6. The subject experiences a drug-related serious adverse event or drug-related severe adverse event. AEs will be considered as drug-related unless clearly unrelated (e.g. events prior to administration of study drug), see Section 5.1.5.1.6.

In addition to these criteria, the investigator may discontinue subjects at any time based on his or her clinical judgment.

Even if the trial treatment is discontinued, the subject remains in the trial and, given his/her agreement, will undergo the procedures for early treatment discontinuation and follow up as outlined in the Flow Chart and Section 6.2.3.

#### 3.3.4.2 Withdrawal of consent to trial participation

Subjects may withdraw their consent to trial participation at any time without the need to justify the decision. If a subject wants to withdraw consent, the investigator should be involved in the discussion with the subject and explain the difference between trial treatment discontinuation and withdrawal of consent to trial participation, as well as explain the options for continued follow up after trial treatment discontinuation, please see Section 3.3.4.1 above

#### 3.3.4.3 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial at any time for any of the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular trial site
- 2. New toxicological findings, serious adverse events, or any safety information invalidating the earlier positive benefit-risk-assessment. More specifically, the trial will be terminated or suspended if more than 50% of the subjects have drug-related and clinically relevant adverse events of moderate or severe intensity, if more than two subjects have drug-related non-serious adverse events of severe intensity or if at least 1 drug-related serious adverse event is reported. AEs will be considered as drug-related unless clearly unrelated (e.g., events prior to administration of study drug), see Section 5.1.5.1.6.

  Any further dosing is only possible after an analysis and evaluation of the harm, review of

Boehringer Ingelheim BI Trial No.: 1405-0007 c24401085-02

**22 November 2018** 

Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

the risk-benefit analysis, submission of a substantial amendment for further dosage and approval by the competent authority and ethics committee.

- 3. Violation of GCP or the CTP impairing the appropriate conduct of the trial-
- 4. The sponsor decides to discontinue the further development of the investigational product

#### 3.3.5 Replacement of subjects

Subjects withdrawn due to drug related adverse events will not be replaced. In case some subjects do not complete the trial for any other reason, the Trial Clinical Monitor together with the Trial Pharmacokineticist and the Trial Statistician are to decide, if and how many subjects will be replaced. A replacement subject will be assigned a unique trial subject number, and will be assigned to the same treatment as the subject replaces.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. TREATMENTS

#### 4.1 INVESTIGATIONAL TREATMENTS

The investigational product has been manufactured by BI Pharma GmbH & Co. KG.

#### 4.1.1 Identity of the Investigational Medicinal Products

The characteristics of the test product are given below:

Substance: BI 1323495

Pharmaceutical formulation: Tablet, film-coated

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength:

Posology: 2-0-0 Route of administration: oral

Duration of use: single dose in treatment T and R

#### 4.1.2 Selection of doses in the trial and dose modifications

In the ongoing first in man trial (1405-0001) it is planned to investigate single doses up to BI 1323495. In this food effect trial, it is intended to administer two single doses of BI 1323495. This dose has been chosen as it corresponds to the assumed therapeutic dose (see Section 1.2.2).

The investigator in this trial 1405-0007 will be informed by the sponsor in writing about the outcome of the documented safety review meeting scheduled after completion of the dose group in trial 1405-0001.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Based on the experience gained during trial 1405-0001, a lower dose of BI 1323495 may be tested in this trial. If the lower dose is selected for safety reasons, this will be implemented via substantial amendment only.

#### 4.1.3 Method of assigning subjects to treatment groups

The randomisation list will be provided to the trial site in advance.

Subjects will be allocated to treatment sequences prior to the first administration of trial medication in the morning of Day 1 (Visit 2). For this purpose, numbers of the randomisation list will be allocated to the subjects by drawing lots. Subjects are then assigned to a treatment sequence according to the randomisation list.

Once a subject number has been assigned, it cannot be reassigned to any other subject.

All subjects may be treated in one cohort, i.e. all subjects may receive treatment on the same calendar day. In case this is not feasible (e.g., due to logistical or recruitment reasons), the group may be split into several cohorts as required. Treatment of all subjects on the same calendar day is acceptable (for safety margin to exposure reached in SRD trial 1405-0001 and for discussion of study-associated risks and safety measures, see Section 1.4).

The randomisation procedure is described in Section <u>7.6</u>.

#### 4.1.4 Drug assignment and administration of doses for each subject

This trial is a 2-way crossover study. All subjects will receive the 2 treatments in randomised order. The treatments to be evaluated are outlined in Table 4.1.4: 1 below.

Table 4.1.4: 1 Dosage and treatment schedule

| Treatment | Substance | Formulation | Unit strength | Dosage | | Total dose |
|---|---|---|---|---|---|---|
| T (Test) | BI 1323495 | Tablet, film-<br>coated | | fed state | as single dose, | |
| R (Reference) | BI 1323495 | Tablet, film-<br>coated | | fasted state | as single dose, | |

Administration of trial medication will be performed after subjects have fasted overnight; fasting is to start no later than 10 h before the scheduled dosing.

In treatment T, a high-fat, high-calorie meal will be served within 30 min before drug administration. The subjects must completely consume the meal prior to drug intake. The composition of the standard high-fat, high-calorie meal is detailed in Table 4.1.4: 2; this meal is in compliance with the FDA guidance 'Food-Effect Bioavailability and Fed Bioequivalence Studies' (R03-2269). For restrictions with regard to diet, see Section 4.2.2.2.

Table 4.1.4: 2 Composition of the high-fat, high-calorie meal

| Ingredients | kcal |
|---------------------------------------------------|------|
| 2 chicken eggs (whole content) for scrambled eggs | 192 |
| 10 g butter for frying scrambled eggs | 75 |

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Ingredients | kcal |
|----------------------------------------|------|
| 35 g fried bacon | 186 |
| 2 toasted slices of wheat bread | 130 |
| 15 g butter for buttering toast slices | 113 |
| 115 g hash brown potatoes | 132 |
| 240 mL whole milk (3.5% fat) | 156 |
| Sum <sup>1</sup> | 984 |

The total caloric content was supplied approximately as following: 150 kcal as protein, 250 kcal as carbohydrate, and 500 to 600 kcal as fat.

The investigator (or authorised designee) will administer the trial medication as an oral dose together with about 240 mL of water to subjects who are in a standing position. For drug administration, the so-called four-eye principle (two-person rule) should be applied. For this, one authorised employee of the trial site should witness the administration of trial medication, and – if applicable – its preparation (e.g. reconstitution), if correct dosage cannot be ensured otherwise.

Subjects will be kept under close medical surveillance until 24 h after drug administration. During the first 4 h after drug administration, subjects are not allowed to lie down (i.e. no declination of the upper body of more than 45 degrees from upright posture).

The treatments will be separated by a wash-out phase of at least 6 days.

# 4.1.5 Blinding and procedures for unblinding

This Phase I trial will be handled in an open fashion throughout (that is, during the conduct, including data cleaning and preparation of the analysis). This is considered acceptable because the potential for bias seems to be low and does not outweigh practical considerations.

Emergency envelopes will not be provided, because the dose of trial medication is known to investigators and subjects.

PK samples will be labelled in such a way that treatment allocation cannot be derived by the analytical site.

#### 4.1.6 Packaging, labelling, and re-supply

The investigational medicinal products will be provided by BI. They will be packaged and labelled in accordance with local law and the principles of Good Manufacturing Practice.

For details of packing and the description of the label, refer to the ISF.

The telephone number of the sponsor and the name, address and telephone number of the trial site are provided in the subject information form. The EudraCT number is indicated on the title page of this protocol as well as on the subject information and informed consent forms.

No re-supply is planned.

c24401085-02

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area in accordance with the recommended (labelled) storage conditions. If necessary, a temperature log must be maintained to make certain that the drug supplies are stored at the correct temperature. If the storage conditions are found to be outside the specified range, the local clinical monitor (as provided in the list of contacts) is to be contacted immediately.

#### 4.1.8 Drug accountability

The investigator or designee will receive the investigational drugs delivered from the sponsor following requirements are fulfilled:

- Approval of the clinical trial protocol by the IRB / ethics committee
- Approval/notification of the regulatory authority, e.g. competent authority
- Availability of the *curriculum vitae* of the Principal Investigator
- Availability of a signed and dated clinical trial protocol

Only authorised personnel documented in the form 'Trial Staff List' may dispense medication to trial subjects. The trial medication must be administered in the manner specified in the CTP.

The investigator or designee must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each subject, and the disposal of unused products. These records will include dates, quantities, batch / serial numbers, expiry ('use-by') dates, and the unique code numbers assigned to the investigational medicinal product and trial subjects. The investigator or designee will maintain records that document adequately that the subjects were provided the doses specified by the CTP and reconcile all investigational medicinal products received from the sponsor. At the time of disposal of remaining trial medication, the investigator or designee must verify that no remaining supplies are in the investigator's possession.

All unused medication will be disposed of locally by the trial site upon written authorisation of the trial clinical monitor. Receipt, usage and disposal of trial medication must be documented on the appropriate forms. Account must be given for any discrepancies.

# 4.2 OTHER TREATMENTS, EMERGENCY PROCEDURES, RESTRICTIONS

#### 4.2.1 Other treatments and emergency procedures

There are no special emergency procedures to be followed. No additional treatment is planned. However, if adverse events require treatment, the investigator can authorise symptomatic therapy. In those cases, subjects will be treated as necessary and, if required, kept under supervision at the trial site or transferred to a hospital until all results of medical evaluations are acceptable.

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.2.2 Restrictions

c24401085-02

#### 4.2.2.1 Restrictions regarding concomitant treatment

In principle, no concomitant therapy is allowed. All concomitant or rescue therapies will be recorded (including time of intake on study days) on the appropriate pages of the CRF.

Acetylsalicylic acid or other drugs that may inhibit platelet aggregation or coagulation should be avoided during the entire study. If necessary, short term use of ibuprofen or paracetamol is acceptable.

## 4.2.2.2 Restrictions on diet and life style

While admitted to the trial site, the subjects will be instructed not to consume any foods or drinks other than those provided by the staff. Standardised meals will be served at the times indicated in the Flow Chart. No food is allowed for at least 4 h after drug intake.

From 1 h before drug intake until lunch, fluid intake is restricted to the milk served with breakfast (see Table 4.1.4: 2), the water administered with the drug, and an additional 240 mL of water at 2 h and 4 h post-dose (mandatory for all subjects). From lunch until 24 h post-dose, total fluid intake is restricted to 3000 mL.

Alcoholic beverages, grapefruits, Seville oranges (sour or bitter oranges) and their juices, and dietary supplements and products containing St. John's wort (*Hypericum perforatum*) are not permitted from 7 days before the first administration of trial medication until after the last PK sample is collected.

Smoking as well as methylxanthine-containing drinks or foods (such as coffee, tea, cola, energy drinks, or chocolate) are not allowed during in-house confinement.

Excessive physical activity (such as competitive sport) should be avoided from 7 days before the first administration of trial medication until the end of trial examination.

Direct exposure to the sun or exposure to solarium radiation should be avoided during the entire study.

#### 4.3 TREATMENT COMPLIANCE

Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

Subjects who are non-compliant (for instance, who do not appear for scheduled visits or violate trial restrictions) may be removed from the trial and the CRF will be completed accordingly (for further procedures, please see Section 3.3.4.1).

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5. ASSESSMENTS

#### 5.1 ASSESSMENT OF SAFETY

#### 5.1.1 Physical examination

At screening, the medical examination will include demographics, height and body weight, smoking and alcohol history (results of smoking and alcohol history not mandatory to be entered into CRF or to be reported), relevant medical history and concomitant therapy, review of inclusion and exclusion criteria, review of vital signs (BP, PR), 12-lead ECG, laboratory tests, and a physical examination. At the end of trial examination, it will include review of vital signs, 12-lead ECG, laboratory tests, and a physical examination.

# 5.1.2 Vital signs

Systolic and diastolic blood pressures (BP) as well as pulse rate (PR) or heart rate (heart rate is considered to be equal to pulse rate) will be measured by a blood pressure monitor (Dinamap Pro 100, GE Medical Systems, Freiburg, Germany) at the times indicated in the Flow Chart, after subjects have rested for at least 5 min in a supine position. All recordings should be made using the same type of blood pressure recording instrument on the same arm, if possible.

#### **5.1.3** Safety laboratory parameters

For the assessment of laboratory parameters, blood and urine samples will be collected by the trial site at the times indicated in the <u>Flow Chart</u> after the subjects have fasted for at least 10 h. For retests, at the discretion of the investigator or designee, overnight fasting is not required.

The parameters that will be determined are listed in Tables 5.1.3:1 and 5.1.3:2. Reference ranges will be provided in the ISF, Section 10.

Manual differential white blood cell count or urine sediment examinations will only be performed if there is an abnormality in the automatic blood cell count or in the urinalysis, respectively.

c24401085-02

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.1.3: 1 Routine laboratory tests

| Functional lab group | BI test name [comment/abbreviation] | A | В | С |
|---|---|---|---|---|
| Haematology | Haematocrit | X | X | X |
| | Haemoglobin | X | X | X |
| | Red Blood Cell Count/Erythrocytes | X | X | X |
| | White Blood Cells/Leucocytes | X | X | X |
| | Platelet Count/Thrombocytes (quant) | X | X | X |
| Automatic WBC | Neutrophils/Leukocytes; Eosinophils/Leukocytes; Basophils/ | X | X | X |
| differential, relative | Leukocytes; Monocytes/Leukocytes; | | | |
| | Lymphocytes/Leukocytes | | | |
| Automatic WBC | Neutrophil, absol.; Eosinophils, absol.; Basophils, absol.; | X | 37 | v |
| differential, absolute | Monocytes, absol.; Lymphocytes, absol. | A | X | X |
| Manual differential | Neut. Poly (segs); Neut. Poly (segs), absol.; Neutrophils | $X^1$ | $X^1$ | $X^1$ |
| WBC (if automatic | Bands; Neutrophils Bands, absol.; Eosinophils/Leukocytes; | | | |
| differential WBC is | Eosinophils, absol.; Basophils/ Leukocytes; Basophils, absol.; | | | |
| abnormal) | Monocytes/ Leukocytes; Monocytes, absol.; | | | |
| , | Lymphocytes/Leukocytes; Lymphocytes, absol. | | | |
| Coagulation | Activated Partial Thromboplastin Time | X | X | X |
| | Prothrombin time – INR (International Normalization Ratio) | X | X | X |
| | Fibrinogen | X | X | X |
| Enzymes | AST [Aspartate transaminase] /GOT, SGOT | X | X | X |
| | ALT [Alanine transaminase] /GPT, SGPT | X | X | X |
| | Alkaline Phosphatase | X | X | X |
| | Gamma-Glutamyl Transferase | X | X | X |
| | Creatine Kinase [CK] | X | X | X |
| | Creatine Kinase Isoenzyme MB [only if CK is elevated] | X | X | X |
| | Lactic Dehydrogenase | X | X | X |
| | Lipase | X | X | X |
| Hormones | Thyroid Stimulating Hormone | X | | |
| Substrates | Glucose (Plasma) | X | X | X |
| | Creatinine | X | X | X |
| | GFR/ CKD-EPI <sup>2</sup> | X | X | X |
| | Bilirubin, Total | X | X | X |
| | Bilirubin, Direct | X | X | X |
| | Protein, Total | X | X | X |
| | Albumin | X | | X |
| | C-Reactive Protein (Quant) | X | X | X |
| | Uric Acid | X | | X |
| | Cholesterol, total | X | | X |
| | Triglyceride | X | | X |
| Electrolytes | Sodium | X | X | X |
| | Potassium | X | X | X |

<sup>&</sup>lt;sup>1</sup> if automatic differential WBC is abnormal

<sup>&</sup>lt;sup>2</sup> estimated glomerular filtration rate according to CKD-EPI formula (<u>R12-1392</u>)

A: parameters to be determined at Visit 1 (screening examination)

B: parameters to be determined at Visits 2 and 3 (for time points refer to Flow Chart)

C: parameters to be determined at Visit 4 (end of trial examination)

Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.1.3: 1 Routine laboratory tests (cont.)

| Functional lab group | BI test name [comment/abbreviation] | A | В | С |
|---|---|---|---|---|
| Urinalysis (Stix) | Urine Nitrite (qual) | X | 1 | X |
| | Urine Protein (qual) | X | | X |
| | Urine Glucose (qual) | X | | X |
| | Urine Ketone (qual) | X | | X |
| | Urobilinogen (qual) | X | | X |
| | Urine Bilirubin (qual) | X | | X |
| | Urine RBC/Erythrocytes (qual) | X | | X |
| | Urine WBC/Leucocytes (qual) | X | | X |
| | Urine pH | X | | X |
| Urine sediment <sup>3</sup> | Only positive findings will be reported (for instance, the | $X^3$ | | $X^3$ |
| (microscopic | presence of sediment bacteria, casts in sediment, squamous | | | |
| examination if | epithelial cells, erythrocytes, leukocytes) | | | |
| erythrocytes, | | | | |
| leukocytes nitrite or | | | | |
| protein are abnormal | | | | |
| in urine) | | | | |

<sup>&</sup>lt;sup>3</sup> if erythrocytes, leukocytes nitrite or protein are abnormal in urinalysis

The tests listed in Table <u>5.1.3: 2</u> are exclusionary laboratory tests that may be repeated as required. The results will not be entered in the CRF/database and will not be reported in the CTR. Except for drug screening, it is planned to perform these tests during screening only. Drug screening will be performed at screening and prior to each treatment period.

Table 5.1.3: 2 Exclusionary laboratory tests

| Functional lab group | Test name |
|-----------------------------|-------------------------------------------|
| Drug screening (urine) | Amphetamine/MDA |
| | Barbiturates |
| | Benzodiazepine |
| | Cannabis |
| | Cocaine |
| | Methadone |
| | Methamphetamines/MDMA/XTC |
| | Opiates |
| | Phencyclidine |
| | Tricyclic antidepressants |
| Infectious serology (blood) | Hepatitis B surface antigen (qualitative) |
| | Hepatitis B core antibody (qualitative) |
| | Hepatitis C antibodies (qualitative) |
| | 1 1 |
| | HIV-1 and HIV-2 antibody (qualitative) |

To encourage compliance with alcoholic restrictions, a breath alcohol test (e.g. Alcotest<sup>®</sup> 7410, Dräger AG, Lübeck, Germany) will be performed prior to each treatment period, and

A: parameters to be determined at Visit 1 (screening examination)

B: parameters to be determined at Visits 2 and 3 (for time points refer to Flow Chart)

C: parameters to be determined at Visit 4 (end of trial examination)
c24401085-02

Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

may be repeated at any time during the study at the discretion of an investigator or designee. The results will not be included in the CTR.

The laboratory tests listed in Tables 5.1.3: 1 and 5.1.3: 2 will be performed

with the exception of

drug screening tests. These tests will be performed at the trial site using M-10/14-PDT test or a comparable test system.

Laboratory data will be transmitted electronically from the laboratory to the trial site.

# 5.1.4 Electrocardiogram

Twelve-lead ECGs (I, II, III, aVR, aVL, aVF, V1 - V6) will be recorded using a computerised electrocardiograph (CardioSoft EKG System, GE Medical Systems, Freiburg, Germany) at the times provided in the Flow Chart.

To achieve a stable heart rate at rest and to assure high quality recordings, the site personnel will be instructed to assure a relaxed and quiet environment, so that all subjects are at complete rest.

All ECGs will be recorded for 10 sec duration after subjects have rested for at least 5 min in a supine position. ECG assessment will always precede all other study procedures scheduled for the same time to avoid compromising ECG quality.

All ECGs will be stored electronically on the Muse CV Cardiology System (GE Medical Systems, Freiburg, Germany). Electrode placement will be performed according to the method of Wilson, Goldberger and Einthoven modified by Mason and Likar (hips and shoulders instead of ankles and wrists).

All locally printed ECGs will be evaluated by the investigator or a designee. Abnormal findings will be reported as AEs (during the trial) or baseline conditions (at screening) if assessed to be clinically relevant by the investigator. Any ECG abnormalities will be carefully monitored and, if necessary, the subject will be removed from the trial and will receive the appropriate medical treatment.

ECGs may be repeated for quality reasons (for instance, due to alternating current artefacts, muscle movements, or electrode dislocation) and the repeated ECG will be used for analysis. Additional (unscheduled) ECGs may be collected by the investigator for safety reasons.

#### 5.1.5 Assessment of adverse events

#### 5.1.5.1 Definitions of adverse events

#### 5.1.5.1.1 Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The following should also be recorded as an AE in the CRF and BI SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination, and laboratory test results, if they are judged clinically relevant by the investigator

If such abnormalities already pre-exist prior to trial inclusion, they will be considered as baseline conditions and should be collected in the eCRF only.

#### 5.1.5.1.2 Serious adverse event

A serious adverse event (SAE) is defined as any AE which fulfils at least one of the following criteria:

- Results in death
- Is life-threatening, which refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe
- Requires inpatient hospitalisation
- Requires prolongation of existing hospitalisation
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly/birth defect
- Is deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse

#### 5.1.5.1.3 AEs considered 'Always Serious'

Cancers of new histology and exacerbations of existing cancer must be classified as a serious event regardless of the time since discontinuation of the trial medication and must be reported as described in <u>5.1.5.2</u>, subsections 'AE Collection' and 'AE reporting to sponsor and timelines'.

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of further AEs, which, by their nature, can always be considered to be 'serious' even though they may not have met the criteria of an SAE as defined above.

The latest list of 'Always Serious AEs' can be found in the eDC system, an electronic data capture system which allows the entry of trial data at the trial site. These events should always be reported as SAEs as described above.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.1.5.1.4 Adverse events of special interest

The term adverse events of special interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESIs need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAEs, please see Section 5.1.5.2.2.

The following are considered as AESIs:

## • Hepatic injury

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, or
- o Aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

These lab findings constitute a hepatic injury alert and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

#### 5.1.5.1.5 Intensity (severity) of AEs

The intensity (severity) of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) that is/are easily tolerated Moderate: Sufficient discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

#### 5.1.5.1.6 Causal relationship of AEs

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by or attributed to the drug class
- A plausible time to onset of the event relative to the time of drug exposure


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Evidence that the event is reproducible when the drug is re-introduced
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications)
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome)
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is reduced)

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned)
- Disappearance of the event even though the trial drug treatment continues or remains unchanged

#### 5.1.5.2 Adverse event collection and reporting

#### 5.1.5.2.1 AE collection

Upon enrolment into a trial, the subject's baseline condition is assessed (for instance, by documentation of medical history/concomitant diagnoses), and relevant changes from baseline are noted subsequently.

Subjects will be required to report spontaneously any AEs as well as the time of onset, end time, and intensity of these events. In addition, each subject will be regularly assessed by the medical staff throughout the clinical trial and whenever the investigator deems necessary. As a minimum, subjects will be questioned for AEs (and concomitant therapies) at the time points indicated in the <u>Flow Chart</u>. Assessment will be made using non-specific questions such as 'How do you feel?'. Specific questions will be asked wherever necessary in order to more precisely describe an AE.

A carefully written record of all AEs shall be kept by the investigator in charge of the trial. Records of AEs shall include data on the time of onset, end time, intensity of the event, and any treatment or action required for the event and its outcome.

The following must be collected and documented on the appropriate CRF(s) by the investigator:

• From signing the informed consent onwards until an individual subject's end of trial:


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- All AEs (serious and non-serious) and all AESIs
- The only exception to this rule are AEs (serious and non-serious) and AESIs in Phase I trials in healthy volunteers, when subjects discontinue from the trial due to screening failures prior to administration of any trial medication. In these cases, the subjects' data must be collected at trial site but will not be entered in the CRF or trial database and will not be reported in the CTR.
- After the individual subject's end of trial:
  - The investigator does not need to actively monitor the subject for AEs but should only report any occurrence of cancer and related SAEs and related AESIs of which the investigator may become aware of by any means of communication, e.g. phone call. Those AEs should, however, not be reported in the CRF.

#### AE reporting to the sponsor and timelines 5.1.5.2.2

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form via fax immediately (within 24 hours) to the sponsor's unique entry point (country specific contact details will be provided in the ISF). The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and fax the BI SAE form.

With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information, the same rules and timeline apply as for initial information.

#### 5.1.5.2.3 Information required

All (S)AEs, including those persisting after the individual subject's end of trial, must be followed up until they have resolved, have been sufficiently assessed as 'chronic' or 'stable', or no further information can be obtained.

#### 5.1.5.2.4 Pregnancy

Once the male subject has been enrolled in the clinical trial and has taken trial medication, and if a partner of the male trial participant becomes pregnant, the investigator must report any drug exposure during pregnancy in a partner of the male trial participant immediately (within 24 hours) by means of Part A of the Pregnancy Monitoring Form to the sponsor's unique entry point, after a written consent of the pregnant partner.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Trials (Part B).

The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and Part B) as well as non-trial specific information and consent for the pregnant partner.

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE and/or AESI, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE form c24401085-02


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

is to be completed. If there is an SAE and/or AESI associated with the pregnancy, an SAE form must be completed in addition.

# 5.2 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

## **5.2.1** Assessment of pharmacokinetics

For the assessment of pharmacokinetics, blood samples will be collected at the time points indicated in the <u>Flow Chart</u>. The actual sampling times will be recorded and used for determination of pharmacokinetic parameters.

#### 5.2.2 Methods of sample collection

#### 5.2.2.1 Blood sampling for pharmacokinetic analysis

For quantification of BI 1323495 concentrations in plasma, 2.7 mL of blood will be drawn from an antecubital or forearm vein into a K2-EDTA (dipotassium ethylenediaminetetraacetic acid)-anticoagulant blood drawing tube at the times indicated in the <u>Flow Chart</u>. Blood will be withdrawn by means of either an indwelling venous catheter or by venepuncture with a metal needle.

The EDTA-anticoagulated blood samples will be centrifuged for approximately 10 min at approximately 2000 x g to 4000 x g and at 4 to 8 °C. Two plasma aliquots will be obtained and stored in polypropylene tubes. The first aliquot should contain at least 0.5 mL of plasma. The process from blood collection until transfer of plasma aliquots into the freezer should be completed within 60 min, with interim storage of blood samples at room temperature. The time each aliquot was placed in the freezer will be documented. Until transfer on dry ice to the analytical laboratory, the aliquots will be stored upright at approximately -20°C or below at the trial site. The second aliquot will be transferred to the analytical laboratory after the bioanalyst has acknowledged safe arrival of the first aliquot. At the analytical laboratory, the plasma samples will be stored at approximately -20°C or below until analysis.

At a minimum, the sample tube labels should list BI trial number, subject number, visit, and planned sampling time.

After completion of the trial, the plasma samples may be used for further methodological investigations (e.g. for stability testing or assessment of metabolites. However, only data related to the analyte and/or its metabolite(s) including anti-drug antibodies (if applicable) will be generated by these additional investigations. The study samples will be discarded after completion of the additional investigations but not later than 5 years after the CTR is archived.

#### **5.2.3** Analytical determinations

BI 1323495 concentrations in plasma will be determined by a validated LC-MS/MS (liquid chromatography tandem mass spectrometry) assay. All details of the analytical method will be available prior to the start of sample analysis.

Boehringer Ingelheim BI Trial No.: 1405-0007

c24401085-02

**22 November 2018** 

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

During sample analysis, the bioanalyst will be blinded to subject allocation and will have no access to the randomisation code.

## 5.2.4 Pharmacokinetic - pharmacodynamic relationship

No analysis of the relationship between pharmacokinetic and pharmacodynamic parameters is planned for this trial.

#### 5.3 BIOBANKING

Not applicable.

#### 5.4 OTHER ASSESSMENTS

# 5.4.1 Pharmacogenomic evaluation

#### 5.5 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements and will be performed in order to monitor subjects' safety and to determine pharmacokinetic parameters in an appropriate way. The scheduled measurements will allow monitoring of changes in vital signs, standard laboratory values, and ECG parameters that might occur as a result of administration of trial medication. The safety assessments are standard, are accepted for evaluation of safety and tolerability of an orally administered drug, and are widely used in clinical trials. The pharmacokinetic parameters and measurements outlined in Section 5.3 are generally used assessments of drug exposure.


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. **INVESTIGATIONAL PLAN**

#### 6.1 VISIT SCHEDULE

Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening, for measurements and assessments scheduled to occur 'before' trial medication administration on Day 1, and the end of trial examination are provided in the Flow Chart.

The acceptable deviation from the scheduled time for vital signs, ECG and laboratory tests will be  $\pm$  15 min for the first 4 h after trial drug administration and  $\pm$  30 min thereafter. Starting from 48 h post administration a deviation from the scheduled time for vital signs, ECG and laboratory tests of  $\pm 120$  min is acceptable.

If scheduled in the Flow Chart at the same time as a meal, blood sampling, vital signs, and 12-lead ECG recordings have to be done first. Furthermore, if several measurements including venepuncture are scheduled for the same time, venepuncture should be the last of the measurements due to its inconvenience to the subject and possible influence on physiological parameters.

For planned blood sampling times, refer to the Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for the determination of pharmacokinetic parameters.

If a subject misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Report Planning Meeting.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening

After having been informed about the trial, all subjects will provide written informed consent in accordance with GCP and local legislation prior to enrolment in the study.

For information regarding laboratory tests (including drug and virus screening), ECG, vital signs, and physical examination, refer to Sections 5.1.1 to 5.1.4.

#### 6.2.2 **Treatment periods**

Each subject is expected to participate in 2 treatment periods (Days -1, 1, 2, 3, 4 and 5 in each period). In addition, an ambulatory visit will be necessary within 3 days prior to the first study drug administration for safety laboratory. At least 6 days will separate drug administrations in the first and second treatment periods.

In the evening of Day -1 of each treatment period, study participants will be admitted to the trial site and kept under close medical surveillance for at least 24 h following drug

Boehringer Ingelheim BI Trial No.: 1405-0007 c24401085-02

**22 November 2018** 

Trial Protocol 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

administration. The subjects will then be allowed to leave the trial site after formal assessment and confirmation of their fitness. All following trial assessments will be performed in an ambulatory fashion.

For details on time points and procedures for collection of plasma samples for PK analysis, refer to Flow Chart and Section 5.2.2.

The safety measurements performed during the treatment period are specified in Section <u>5.1</u> of this protocol and in the <u>Flow Chart</u>. For details on times of all other trial procedures, refer to the <u>Flow Chart</u>. AEs and concomitant therapy will be assessed continuously from screening until the end of trial examination.

#### 6.2.3 Follow-up period and trial completion

For AE assessment, laboratory tests, recording of ECG and vital signs, and physical examination during the follow-up period, see Section <u>5.1</u>.

Subjects who discontinue treatment before the end of the planned treatment period should undergo the EoTrial Visit.

All abnormal values (including laboratory parameters) that are assessed as clinically relevant by the investigator will be monitored using the appropriate tests until a return to a medically acceptable level is achieved. (S)AEs persisting after a subject's EoTrial Visit must be followed until they have resolved, have been sufficiently characterised, or no further information can be obtained.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN – MODEL

The main objective of this trial is to investigate the relative bioavailability of BI 1323495 administered as tablet formulation in the fed state (Test, T) compared to BI 1323495 administered as tablet formulation in the fasted state (Reference, R) on the basis of the primary and secondary pharmacokinetic endpoints, as listed in Section 2.1.2 and 2.1.3. The trial is designed to allow intra-subject comparisons and will be evaluated statistically by use of a linear model for logarithmically transformed PK endpoints.

A further objective is to evaluate and compare further pharmacokinetic parameters between the treatments. These pharmacokinetic parameters will be assessed by descriptive statistics.

The assessment of safety and tolerability is a further objective of this trial, and will be evaluated by descriptive statistics for the parameters specified in Section 2.2.2.2.

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

The relative bioavailability of BI 1323495 under fed and fasted conditions will be estimated by the ratios of the geometric means (test/reference), and their corresponding 2-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at the 5% significance level. Since the main focus is on estimation and

#### 7.3 PLANNED ANALYSES

#### Analysis sets

Statistical analyses will be based on the following analysis sets:

- Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of study drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model based analyses of PK parameters will be based on the PKS.

Adherence to the protocol will be assessed by the trial team. Important protocol violation (IPV) categories will be suggested in the TSAP, IPVs will be identified no later than in the Report Planning Meeting, and the IPV categories will be updated as needed.


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Pharmacokinetics

The pharmacokinetic parameters listed in Section 2.1 for BI 1323495 will be calculated according to the relevant Standard Operating Procedure (SOP) of the Sponsor

Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol violation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol violations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Use of restricted medications

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- The subject experienced emesis that occurred at or before two times median t<sub>max</sub> of the respective treatment (Median t<sub>max</sub> is to be determined excluding the subjects experiencing emesis)
- A predose concentration is >5% C<sub>max</sub> value of that subject
- Missing samples/concentration data at important phases of PK disposition curve

Plasma concentration data and parameters of a subject which is flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses. Descriptive and inferential statistics of PK parameters will be based on the PKS.

Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of pharmacokinetic parameters. Concentrations used in the pharmacokinetic calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).

# 7.3.1 Primary endpoint analyses

#### Primary analyses

The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' will be considered as random, whereas the other effects will be considered as fixed. The model is described by the following equation:

$$y_{ijkm} = \mu + \zeta_i + s_{im} + \pi_i + \tau_k + e_{ijkm}$$
, where

 $y_{ijkm}$  = logarithm of response measured on subject m in sequence i receiving treatment

c24401085-02 Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

k in period j,

 $\mu =$  the overall mean,

 $\zeta_i$  = the i<sup>th</sup> sequence effect, i = 1, 2,

 $s_{im}$  = the effect associated with the m<sup>th</sup> subject in the i<sup>th</sup> sequence, m = 1, 2,...,6

 $\pi_i$  = the j<sup>th</sup> period effect, j = 1, 2,

 $\tau_k =$  the  $k^{th}$  treatment effect, k = 1, 2,

e<sub>ijkm</sub> = the random error associated with the m<sup>th</sup> subject in sequence i who received treatment k in period j.

where  $s_{im} \sim N(0, \sigma_B^2)$  i.i.d.,  $e_{ijkm} \sim N(0, \sigma_W^2)$  i.i.d. and  $s_{im}$ ,  $e_{ijkm}$  are independent random variables.

Point estimates for the ratios of the geometric means (test/reference) for the primary endpoints (see Section 2.1) and their two-sided 90% confidence intervals (CIs) will be provided.

For each endpoint, the difference between the expected means for log(T)-log(R) will be estimated by the difference in the corresponding adjusted means (Least Squares Means). Additionally their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

## Further exploratory analyses

The same statistical model as stated above will be repeated for the primary endpoints but with all sources of variation ('sequence', 'subjects within sequences', 'period', 'treatment') considered as fixed effects.

In addition to the model based approach all parameters will be calculated and analysed descriptively.

#### 7.3.2 Secondary endpoint analyses

The secondary endpoints (refer to Section 2.1.3) will be calculated according to the BI SOP 'Standards and processes for analyses performed within Clinical Pharmacokinetics/
Pharmacodynamics' and will be assessed statistically using the same methods as described for the primary endpoints.


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7.3.4 Safety analyses

Safety will be analysed based on the assessments described in Section <u>2.2.2.2</u>. All treated subjects (TS, refer to Section <u>7.3</u>) will be included in the safety analysis. Safety analyses will be descriptive in nature and based on BI standards. No hypothesis testing is planned.

For all analyses, the treatment actually administered (= treatment at onset) to the subject will be used (any deviations from the randomised treatment will be discussed in the minutes of the Report Planning Meeting).

Treatments will be compared in a descriptive way. Tabulations of frequencies/proportions will be used to evaluate categorical (qualitative) data, and tabulations of descriptive statistics will be used to analyse continuous (quantitative) data.

Measurements (such as ECG, vital signs, or laboratory parameters) or AEs will be assigned to treatments (see Section 4.1) based on the actual treatment at the planned time of the measurement or on the recorded time of AE onset (concept of treatment emergent AEs). Therefore, measurements planned or AEs recorded prior to first intake of trial medication will be assigned to the screening period, those between first trial medication intake and end of trial termination date will be assigned to the treatment period. These assignments including the corresponding time intervals will be defined in detail in the TSAP. Note that AEs occurring after the last per protocol contact but entered before final database lock will be reported to Pharmacovigilance only and will not be captured in the trial database.

Additionally, further treatment intervals (analysing treatments) may be defined in the TSAP in order to provide summary statistics for time intervals, such as combined treatments, ontreatment totals, or periods without treatment effects (such as screening and follow-up intervals).

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Frequency, severity, and causal relationship of AEs will be tabulated by treatment, system organ class, and preferred term. SAEs, AESIs (see Section <u>5.2.5.1</u>), and other significant AEs (according to ICH E3) will be listed separately.

Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

Laboratory data will be compared to their reference ranges. Values outside the reference range as well as values defined as possibly clinically significant will be highlighted in the listings. Additionally, differences from baseline will be evaluated.

Vital signs or other safety-relevant data will be assessed with regard to possible on-treatment changes from baseline.

Relevant ECG findings will be reported as AEs.

#### 7.4 INTERIM ANALYSES

No interim analysis is planned.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.5 HANDLING OF MISSING DATA

# **7.5.1** Safety

It is not planned to impute missing values for safety parameters.

#### 7.5.2 Pharmacokinetics

Handling of missing PK data will be performed according to the relevant Corporate Procedure .

PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

#### 7.6 RANDOMISATION

Subjects will be randomised to one of the 2 treatment sequences in a 1:1 ratio. The block size will be documented in the CTR.

The sponsor will arrange for the randomisation as well as packaging and labelling of trial medication. The randomisation list will be generated using a validated system that uses a pseudo-random number generator and a supplied seed number so that the resulting allocation is both reproducible and non-predictable.

The randomisation list will contain additional blocks to allow for subject replacement (refer to Section 3.3.5).

## 7.7 DETERMINATION OF SAMPLE SIZE

It is planned to enter a total of 12 subjects in the trial, because this sample size is considered sufficient to achieve the aims of this exploratory trial.

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY, AND ADMINISTRATIVE STRUCTURE

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU regulation 536/2014, and other relevant regulations. Investigators and site staff must adhere to these principles.

Standard medical care (prophylactic, diagnostic, and therapeutic procedures) remains the responsibility of the subject's treating physician.

The investigator will inform the sponsor immediately of any urgent safety measures taken to protect the trial subjects against any immediate hazard, as well as of any serious breaches of the protocol or of ICH GCP.

The Boehringer Ingelheim transparency and publication policy can be found on the following web page: trials.boehringer-ingelheim.com. As a general rule, no trial results should be published prior to archiving of the CTR.

The terms and conditions of the insurance coverage are made available to the investigator and the subjects, and are stored in the ISF.

## 8.1 TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB / Independent Ethics Committee (IEC and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments. Prior to a subject's participation in the trial, written informed consent must be obtained from each subject (or the subject's legally accepted representative) according to ICH-GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional subject-information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional subject information must be given to each subject or the subject's legally accepted representative.

The subject must be given sufficient time to consider participation in the trial. The investigator or delegate obtains written consent of the subject's own free will with the informed consent form after confirming that the subject understands the contents. The investigator or delegate must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.

Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

The consent and re-consenting process should be properly documented in the source documentation.


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8.2 DATA QUALITY ASSURANCE

A risk-based approach is used for trial quality management. It is initiated by the assessment of critical data and processes for trial subject protection and reliability of the results as well as identification and assessment of associated risks. An Integrated Quality and Risk Management Plan documents the rationale and strategies for risk management during trial conduct including monitoring approaches, vendor management and other processes focusing on areas of greatest risk.

Continuous risk review and assessment may lead to adjustments in trial conduct, trial design or monitoring approaches.

A quality assurance audit/inspection of this trial may be conducted by the sponsor, sponsor's designees, or by IRB / IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial..

#### 8.3 RECORDS

CRFs for individual subjects will be provided by the sponsor. For drug accountability, refer to Section 4.1.8.

#### **8.3.1** Source documents

In accordance with regulatory requirements, the investigator should prepare and maintain adequate and accurate source documents and trial records for each trial subject that include all observations and other data pertinent to the investigation. Source data as well as reported data should follow the 'ALCOA principles' and be <u>attributable</u>, <u>legible</u>, <u>contemporaneous</u>, original, and accurate. Changes to the data should be traceable (audit trail).

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained.

Before providing any copy of subjects' source documents to the sponsor, the investigator must ensure that all subject identifiers (e.g., subject's name, initials, address, phone number, and social security number) have properly been removed or redacted to ensure subject confidentiality.

If the subject is not compliant with the protocol, any corrective action (e.g. re-training) must be documented in the subject file.

For the CRF, data must be derived from source documents, for example:


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Subject identification: sex, year of birth (in accordance with local laws and regulations)
- Subject participation in the trial (substance, trial number, subject number, date subject was informed)
- Dates of subject's visits, including dispensing of trial medication
- Medical history (including trial indication and concomitant diseases, if applicable)
- Medication history
- AEs and outcome events (onset date [mandatory], and end date [if available])
- SAEs (onset date [mandatory], and end date [if available])
- Concomitant therapy (start date, changes)
- Originals or copies of laboratory results and other imaging or testing results, with proper documented medical evaluation (in validated electronic format, if available)
- ECG results (original or copies of printouts)
- Completion of subject's participation in the trial (end date; in case of premature discontinuation, document the reason for it, if known)
- Prior to allocation of a subject to a treatment into a clinical trial, there must be
  documented evidence in the source data (e.g. medical records) that the trial participant
  meets all inclusion criteria and does not meet any exclusion criteria. The absence of
  records (either medical records, verbal documented feedback of the subject or testing
  conducted specific for a protocol) to support inclusion/exclusion criteria does not
  make the subject eligible for the clinical trial.

#### 8.3.2 Direct access to source data and documents

The investigator /institution will allow site trial-related monitoring, audits, IRB / IEC review and regulatory inspections. Direct access must be provided to the CRF and all source documents/data, including progress notes, copies of laboratory and medical test results, which must be available at all times for review by the Clinical Research Associate, auditor and regulatory inspector (e.g. FDA). They may review all CRFs and informed consents. The accuracy of the data will be verified by direct comparison with the source documents described in Section 8.3.1. The sponsor will also monitor compliance with the protocol and GCP.

#### 8.3.3 Storage period of records

#### Trial site:

The trial site(s) must retain the source and essential documents (including ISF) according to the local requirements valid at the time of the end of the trial.


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Sponsor:

The sponsor must retain the essential documents according to the sponsor's SOPs.

#### 8.4 EXPEDITED REPORTING OF ADVERSE EVENTS

BI is responsible to fulfil their legal and regulatory reporting obligation in accordance with regulatory requirements.

#### 8.5 STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY

Individual subject data obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted in Section 8.7.

Data protection and data security measures are implemented for the collection, storage and processing of patient data in accordance with the principles 6 and 12 of the WHO GCP handbook.

Personalised treatment data may be given to the subject's personal physician or to other appropriate medical personnel responsible for the subject's welfare. Data generated at the site as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

# 8.5.1 Collection, storage and future use of biological samples and corresponding data

Measures are in place to comply with the applicable rules for the collection, storage and future use of biological samples and clinical data, in particular

- Sample and data usage has to be in accordance with the informed consent
- The BI-internal facilities storing biological samples from clinical trial participants as well as the external storage facility are qualified for the storage of biological samples collected in clinical trials.
- An appropriate sample and data management system, incl. audit trail for clinical data and samples to identify and destroy such samples according to ICF is in place
- A fit for the purpose documentation (e.g. biomarker proposal, analysis plan and report) ensures compliant usage
- If applicable, a fit for purpose approach will be used for assay/equipment validation depending on the intended use of the biomarker data

Samples and/or data may be transferred to third parties and other countries as specified in the ICF.

#### 8.6 TRIAL MILESTONES

The start of the trial is defined as the date of the enrolment of the first subject in the trial.

The <u>end of the trial</u> is defined as the 'date of the last visit of the last subject in whole trial' ('Last Subject Completed') or 'end date of the last open AE' or 'date of the last follow-up test' or 'date of an AE has been decided as sufficiently followed-up', whichever is latest.

Boehringer Ingelheim BI Trial No.: 1405-0007 c24401085-02

**22 November 2018** 

#### **Trial Protocol**


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

<u>Early termination of the trial</u> is defined as the premature termination of the trial for any reason before the end of the trial as specified in this protocol.

<u>Temporary halt of the trial</u> is defined as any unplanned interruption of the trial by the sponsor with the intention to resume it.

<u>Suspension of the trial</u> is defined as an interruption of the trial based on a Health Authority request.

The EC/competent authority in each participating EU member state will be notified about the trial milestones according to the laws of each member state.

A final report of the clinical trial data will be written only after all subjects have completed the trial in all countries (EU or non-EU), so that all data can be incorporated and considered in the report.

The sponsor will submit to the EU database a summary of the final trial results within one year from the end of a clinical trial as a whole, regardless of the country of the last patient (EU or non-EU).

#### 8.7 ADMINISTRATIVE STRUCTURE OF THE TRIAL

The trial is sponsored by Boehringer Ingelheim (BI).

The trial will be conducted at the

, under the supervision of the Principal Investigator. Relevant documentation on the participating (Principal) Investigators (e.g. their curricula vitae) will be filed in the ISF.

BI has appointed a Trial Clinical Monitor, responsible for coordinating all required trial activities, in order to

- Manage the trial in accordance with applicable regulations and internal SOPs
- Direct the clinical trial team in the preparation, conduct, and reporting of the trial
- ensure appropriate training and information of local clinical monitors (CML), Clinical Research Associates, and investigators of participating trial sites

The trial medication will be provided by the Clinical Trial Supplies Unit, BI Pharma GmbH & Co. KG, Biberach, Germany.

Safety laboratory tests will be performed by the local laboratory of the trial site

Analyses of BI 1323495 concentrations in plasma will be performed

On-site monitoring will be performed by BI or a contract research organisation appointed by BI.

Data management and statistical evaluation will be done by BI according to BI SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

c24401085-02 Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

| R03-2269 | Guidance for industry: food-effect bioavailability and fed bioequivalence |
|---|---|
| | studies. In: U.S. Department of Health and Human Services, Food and |
| | Drug Administration, Center for Drug Evaluation and Research (CDER) |
| | 2002:1-9. |

R12-1392 Levey AS, Stevens LA, Schmid CH, Zhang Y, Castro AF, Feldman HI, Kusek JW, Eggers P, Lente F van, Greene T, Coresh J, Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI). A new equation to estimate glomerular filtration rate. Ann Intern Med 2009;150(9):604-612.

Boehringer Ingelheim BI Trial No.: 1405-0007 c24401085-02 **22 November 2018** 

Trial Protocol


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

R94-1529 Chow SC, Liu JP. Design and Analysis of Bioavailability and Bioequivalence Studies. New York: Marcel Dekker Inc; 1992.

**Boehringer Ingelheim** BI Trial No.: 1405-0007

c24401085-02

**22 November 2018** 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2 **UNPUBLISHED REFERENCES**

05 Apr 2018. c21238478-01 Investigator's Brochure BI 1323495.

**Trial Protocol** 


**Boehringer Ingelheim** BI Trial No.: 1405-0007

**22 November 2018** 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

#### **APPENDICES 10.**

Not applicable.

c24401085-02


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11. **DESCRIPTION OF GLOBAL AMENDMENT(S)**

#### 11.1 **GLOBAL AMENDMENT 1**

| Date of amendment | | 22 November 2018 | |
|---|---|---|---|
| EudraCT number | | 2018-002792-18 | |
| EU number | | | |
| BI Trial number | | | |
| BI Investigational Medicinal | | BI 1323495 | |
| Product(s) | | | |
| Title of protocol | | Relative bioavailability of BI 1323495 following | |
| _ | | oral administration under fed and fasted conditions | |
| | | in healthy male subjects (an open-label, randomised, | |
| | | single-dose, two-period, two-sequence crossover | |
| | | study) | |
| To be implemented only after approval of the IRB / IEC / Competent | | | |
| Authorities | | | |
| To be implemented immediately in order to eliminate hazard – IRB / IEC / | | | |
| Competent Authority to be no | tified | of change with request for approval | |
| Can be implemented without | IRB/ | IEC / Competent Authority approval as | |
| changes involve logistical or a | dmini | istrative aspects only | |
| Section to be changed | 1 | Flow Chart | |
| | 2 | Section 1.2.4 Clinical experience in humans | |
| | 3 | Section 1.4 Benefit – Risk Assessment | |
| | 4 | Section 3.3.3 Exclusion criteria | |
| | 5 | Section 3.3.4.1 Discontinuation of trial treatme | nt |
| | 6 | Section 3.3.4.3 Discontinuation of the trial by t | the |
| | | sponsor | |
| | | Section 3.3.5 Replacement of subjects | |
| | 8 | Section 4.1.3 Method of assigning subjects to | |
| | treatment groups | | |
| | 9 | Section 5.1.3 Safety laboratory parameters | |
| | 10 Section 5.2.2.1 Blood sampling for pharmacokinetic | | inetic |
| analysis | | analysis | |

c24401085-02

**Trial Protocol** 


Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| D | 1 | DV1:1-1-1-1-1-1-1-1-1-1-1-1-1-1-1- |
|---|---|---|
| Description of change | 1 | PK sampling schedule adapted based on SRD data; |
| | | additional ECG/VS at 2h postdose |
| 2<br>3<br>4<br>5<br>6<br>7<br>8<br>9<br>10 | | Preliminary data from SRD trial 1405-0001 |
| | | amended |
| | | Benefit – risk assessment amended based on data |
| | | gained in SRD trial. |
| | | Exclusion criterion 20 more precisely described |
| | | Additional criterion for individual treatment |
| | | discontinuation introduced. |
| | | Discontinuation of the trial by the sponsor, point 2 |
| | | clarified by more detailed description. |
| | | Clarification: subjects withdrawn for drug related |
| | | AEs will not be replaced. |
| | | Explanation that all subjects may be dosed in one |
| | | cohort on the same calendar day. |
| | | Test name of drug screen corrected. |
| | | PK blood samples may be stored at room |
| | | temperature until centrifuged. |
| Rationale for change | 1 | In the SRD trial, maximum plasma concentrations |
| | | were reached earlier than expected based on |
| | | preclinical data; therefore the sampling schedule for |
| | | PK was adapted accordingly |
| | 2/3 | To address request by competent authority / ethics |
| | | committee; to give sound ground for dose selection, |
| | | trial design, and safety measures. |
| | 4 | Clarification requested by ethics committee. |
| | 5 | Addition requested by FDA (protocol was submitted |
| | | to FDA to open IND). |
| | 6 | To address request by competent authority. |
| | 7 | To address request by competent authority. |
| | 8 | Clarification requested by competent authority. |
| | 9 | Name of drug screen test was incorrect. |
| | 10 | Interim storage on ice not necessary according to |
| | 10 | stability data. |
| | | smornly data. |



#### APPROVAL / SIGNATURE PAGE

Document Number: c24401085 Technical Version Number: 2.0

Document Name: clinical-trial-protocol-revision-1

**Title:** Relative bioavailability of BI 1323495 following oral administration under fed and fasted conditions in healthy male subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study)

# **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Author-Trial Statistician | 22 Nov 2018 13:44 CET | |
| Author-Clinical Trial Leader | | 22 Nov 2018 13:51 CET |
| Author-Trial Clinical<br>Pharmacokineticist | 22 Nov 2018 14:14 CET | |
| Approval-Therapeutic Area | | 23 Nov 2018 10:44 CET |
| Approval-Team Member Medicine | 23 Nov 2018 11:39 CET | |
| Verification-Paper Signature<br>Completion | | 26 Nov 2018 09:13 CET |

Boehringer IngelheimPage 2 of 2Document Number: c24401085Technical Version Number: 2.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|